CLINICAL TRIAL: NCT02897037
Title: Bivalirudin vs Heparin During Primary Percutaneous Coronary Intervention in Acute Myocardial Infarction: A Randomised Controlled Trial
Brief Title: Bivalirudin in Acute Myocardial Infarction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bright2
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Acute Myocardial Infarction
Keywords: Bivalirudin; Acute myocardial infarction; percutaneous transluminal coronary angioplasty
MeSH Terms: interventions — bivalirudin; Heparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bivalirudin (Experimental): Bivalirudin will be started in the cath lab, 0.75 mg/kg intravenous bolus followed by 1.75 mg/kg per h infusion; if ACT<225s 5min after bolus, an additional dose of 0.3mg/kg bolus should be given. After procedure, a prolonged infusion (1.75mg/kg per h) will be given for at least 30 min (totally no more than 4 h) followed by a reduced dose infusion (0.2mg/kg per h) up to 20 h.
  Interventions: Drug: Bivalirudin
- Heparin monotherapy (Active Comparator): 100 IU/kg intravenous bolus. If ACT <225s 5 min after bolus injection, additional dose of heparin (20U/kg) will be given.
  Interventions: Drug: heparin

INTERVENTIONS:
Drug: Bivalirudin — Patients would be given anticoagulant therapy with bivalirudin in acute myocardial infarction during emergency PCI operation.
  Other Names: Taijianing
  Arms: Bivalirudin
Drug: heparin — heparin monotherapy
  Other Names: Gansu
  Arms: Heparin monotherapy

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of bivalirudin in AMI patients with DES.

This is a prospective, randomized, single-blind, active drug controlled multicenter clinical research and the study would enrolled a total of 380 AMI patients undergoing percutaneous coronary intervention (PCI) to one of two antithrombotic regimens: bivalirudin alone, or unfractionated heparin alone. All enrolled patients would be followed-up to 30 days.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blind, active drug controlled multicenter clinical research and the study would enrolled a total of 380 AMI patients undergoing percutaneous coronary intervention (PCI) to one of two antithrombotic regimens: bivalirudin alone, or unfractionated heparin alone. All enrolled patients would be followed-up to 30 days. The purpose of the study is to evaluate the efficacy and safety of bivalirudin in AMI patients with DES.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years old
2. Planned emergency PCI for acute myocardial infarction (STEMI) Symptom onset within 12h for STEMI (or within 12-24 hrs for patients have unrelieved chest pain, continuous ST elevation or new developed LBBB)
3. Provide written informed consent.

Exclusion Criteria:

1. Age <18 or >80 years.
2. Any anticoagulant drugs were regularly used within 3 months.
3. Any anticoagulant agents were used 48 h before randomization.
4. Active bleeding or bleeding constitution, bleeding tendency, including the recent retina or vitreous hemorrhage (1 months), GI or urinary tract hemorrhage (3 months), cerebral hemorrhage (6 months) or cerebral infarction history (3 months), etc.
5. Hemoglobin < 90 g/L or platelet count < 100 * 109 / L.
6. Untreated or uncontrolled hypertension > 180/110 mmHg.
7. Elevated ALT level higher than three times of the normal upper limit;severe renal insufficiency (eGFR < 30 mL/min / 1.73 m2).
8. Heparin induced thrombocytopenia.
9. Suspicious aortic dissection, pericarditis and subacute bacterial endocarditis.
10. Known allergy to the study drugs and instruments (UFH, bivalirudin, aspirin and clopidogrel, stainless steel, contrast agents, etc.), or those allergic constitution.
11. Pregnancy , lactation or plan to be pregnant.
12. Known serious progressive diseases such as malignant tumor or prognosis of the patients with severe failure;the survival time < 6 months.
13. Unsuitable for PCI.
14. Attended any clinical trial 1 month before randomised.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Net Adverse Clinical Events | 30 days
  A composite of all cause death, reinfarction, urgent target vessel revascularization, stroke and any bleedings

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) | 30 days
  A composite of all cause death, reinfarction, target vessel revascularization or stroke
Any bleedings (BARC class) | 30 days
  Including all BARC class (class 3-5)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology，General Hospital of Shenyang Military Region, Shanyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided